CLINICAL TRIAL: NCT04624789
Title: Eight At One Stroke: Attention Gangliosidoses A Registry Study for Patients With Gangliosidoses
Brief Title: Registry Gangliosidoses
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: SphinCS Lyso Gemeinnutzige UG (Haftungsbeschrankt) (Other)
Responsible Party: Sponsor
Other Study IDs: D001
Record Dates: First submitted 2020-10-29; First posted 2020-11-12 (Actual); Last update posted 2020-11-12 (Actual); Status verified 2020-10

CONDITIONS: Gangliosidoses; GM1 Gangliosidosis; Morquio B Disease; Sialidosis; Galactosialidosis; Gm2-Gangliosidosis, Variant B1; Tay-Sachs Disease; Sandhoff Disease; GM2 Activator Deficiency
Keywords: Gangliosides; ß-Galactosidase; Neuraminidase; Protective Protein/Cathepsin A; Hexosaminidase A; Hexosamidase A&B; GM2-activator-protein
MeSH Terms: conditions — Gangliosidoses; Gangliosidosis, GM1; Mucopolysaccharidosis IV; Mucolipidoses; Neuraminidase deficiency with beta-galactosidase deficiency; Gm2-Gangliosidosis, Variant B1; Tay-Sachs Disease; Sandhoff Disease; Tay-Sachs Disease, AB Variant; Gangliosidoses, GM2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — DBS Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- GM1-Gangliosidosis - Sialidosis: Confirmed diagnosis of:
  * GM1-Gangliosidosis Morquio B Variant
  * Sialidosis
  * Galactosialidosis
- GM2-Gangliosidoses: Confirmed diagnosis of:
  * Tay-Sachs Disease, incl. B1-Variante
  * Sandhoff Disease
  * GM2-Activator-Deficiency

SUMMARY:
The clinical project "Eight At One Stroke: Attention Gangliosidoses" represents a clinical registry for recording the clinical manifestation and the disease progression of gangliosidoses. The intention of this project is to better understand the manifestation and progression of gangliosidoses and to raise awareness of these disorders in the public health service. The patients or their families, respectively, will be integrated in the study in order to measure Patient Outcome and to objectify the psychosocial burden for the patient and his family. The study has a retrospective and a prospective part. It is planned to transfer the data of the study into a continuous registry.

DETAILED DESCRIPTION:
1. Aim of the Project

   * The aim of the project is to collect fundamental epidemiological and clinical data, such as prevalence and incidence, but also data regarding phenotype, diagnosis and mutation spectrum.
   * To understand the natural course of these diseases seems to be very important for individual advice of families and additionally for planning drug studies.
   * In this study it should also be analyzed how the families and their setting have perceived the disease manifestation. Their perception will be compared to clinical findings and symptoms that were noticed by the physician. The medical history may indicate which symptoms and findings may lead to a well-directed diagnosis.
   * Clinical and genetic data, that also concern aspects of social medicine, of a greater cohort will raise the awareness of pharmaceutical companies that develop new drugs and will increase the chance of patients to participate in a clinical trial.
   * The project will enable validation of biomarkers that may be useful for diagnostic purposes and also for monitoring laboratory parameters during a trial.
   * Patients and their families are involved in the development and procedure of the study. They become a voice and are noticed as partners in the public health service.

3. Background 3.1 Gangliosidoses Gangliosidoses represent autosomal-recessive lysosomal storage disorders, caused by a defect in the lysosomal degradation of gangliosides, resulting in accumulation of these substrates in several organs. Gangliosidoses are divided in eight different diseases according to their biochemical and genetic defect: Four disorders are assigned to GM2-Gangliosidoses, four belong to the Neuraminidase-ß-Galactosidase complex. Gangliosidoses are characterized by more or less pronounced progressive loss of mental and motor capabilities. In patients with a more attenuated phenotype the diagnosis is done often very late, as the typical clinical "classical" features are commonly lacking. Maybe adult patients were never diagnosed.

The diseases result from the accumulation of gangliosides, caused by genetic defects of enzymes or other proteins that are involved in the lysosomal degradation of these complex lipids.

3.2 Classification of Gangliosides GM1-Gangliosidosis - Sialidosis

* GM1-Gangliosidosis (1) Morquio B Variant (2) ß-Galactosidase
* Sialidosis (3) Neuraminidase
* Galactosialidosis (4) Protective Protein/Cathepsin A

GM2-Gangliosidoses

* Tay-Sachs Disease (5), incl. B1-Variante (6) Hexosaminidase A
* Sandhoff Disease (7) Hexosamidase A&B
* GM2-Activator-Deficiency (8) GM2-activator-protein

3.3 Clinical Phenotypes The degree of clinical expression regarding the age of first manifestation, rate of progression and symptoms is extremely heterogeneous and reaches from the lethal hydrops fetalis to the rapidly progressive and to the slowly progressive adult form. The underlying mutations determine the enzyme respectively protein deficiency, in the more attenuated forms, however, the phenotype is additionally influenced by epigenetic factors and the environment. Generally five phenotypic forms are distinguished that differ in the age of first symptoms.

Hydrops fetalis Gangliosidoses can manifest as hydrops fetalis that is defined as fetal fluid accumulation in at least two organ systems, such as ascites, pleural and pericardium effusion and generalized edema. Hydrops fetalis, that mostly leads to intrauterine death, was surprisingly not observed in GM2-gangliosidoses.

Infantile Gangliosidoses Patients with the so-called "classical" infantile form manifest after birth with developmental delay. Between the age of three to six months significant muscular hypotonia becomes obvious. Often, but not exclusively, in GM2-gangliosidoses the parents observe as first symptom an excessive response to an acoustic stimulus with sudden hyperextension of arms and legs and muscle jerks. A cherry-red spot at the eye fundus and a macrocephaly may lead to the diagnosis. A so-called "Hurler-phenotype" is seen in infants with sialidosis, galactosialidosis and GM1-gangliosidoses.

Late-infantile and juvenile Gangliosidoses It is often not possible to differentiate between late.infantile and juvenile gangliosidoses: In young children the parents observe deficits in motor and speech development, later these capabilities get lost. The occurrence of epilpetic seizures implies a bad prognosis. In GM2-gangliosidoses the tetraparesis is hypotonic and floppy, in GM1-gangliosidoses dystonic and spastic. The progressive visual impairment can result in blindness.

Late-onset Gangliosidoses Patients with late-onset (or chronic-adult) type of gangliosidoses present with cerebellar signs such as ataxia, dysarthria and hypotonia. Late-onset GM2-gangliosidoses are characterized by intention tremor and dysmetria, in late-onset GM1-gangliosidoses dystonia and spasticity are the leading neurological symptoms. Prior to the occurrence of neurological symptoms psychoses and episodes of psychosis may appear that later on may dominate the disease manifestation. The cognitive abilities are hardly impaired, due to the severe dysarthria, however, it may be difficult to correctly evaluate the cognitive function. Because in adult gangliosidoses the motor neuron is involved, the patients may resemble individuals with Friedreich-Ataxia ot SMA, for which reason a differentiation between thoMedise disorders may be difficult

ELIGIBILITY:
Inclusion Criteria:

* Biochemically and/or genetically affirmed diagnosis of a gangliosidosis
* The patient or respectively the parents or the caregiver (for children or older underage patients) have given written informed consent

Exclusion Criteria:

* The diagnosis of a gangliosidosis has not biochemically or genetically confirmed.
* A written informed consent of the patient or parents/acaregiver does not exist.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Gangliosidoses
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-06-08 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2025-06-07 (Estimated)

PRIMARY OUTCOMES:
Disease progression will be assessed by the 8 in 1 score | 5 years
  Disease progression was assessed by the 8 in 1 score, which is a disease specific instrument adapted from other scores in neurodegenerative and lysosomal diseases (NPC, CLN). The instrument is designed to monitor disease progession and measure disease severity. The 8 in 1 score summarizes 8 domains (partizipation, medical care, ambulation, manipulation, swallowing, speech, epilepsy and cognition) ranging from 0 - 40. A higher score indicates more severe clinical impairment.

SECONDARY OUTCOMES:
Characterization of the first neurological symptom | 5 years
  In a systematic interview all aspects of medical history and development will be acquisited. The first neurological symptom will be reflected in view of parents/caregiver, GP and disease expert. The timepoint of occurrance and who recognized the finding will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- SphinCS Lyso gemeinnützige UG (haftungsbeschränkt), Hochheim am Main, Hesse, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Harding AE, Young EP, Schon F. Adult onset supranuclear ophthalmoplegia, cerebellar ataxia, and neurogenic proximal muscle weakness in a brother and sister: another hexosaminidase A deficiency syndrome. J Neurol Neurosurg Psychiatry. 1987 Jun;50(6):687-90. doi: 10.1136/jnnp.50.6.687. PMID 2956362
- [Background] Neudorfer O, Kolodny EH. Late-onset Tay-Sachs disease. Isr Med Assoc J. 2004 Feb;6(2):107-11. No abstract available. PMID 14986470
- [Background] Tutor JC. Biochemical characterization of the GM2 gangliosidosis B1 variant. Braz J Med Biol Res. 2004 Jun;37(6):777-83. doi: 10.1590/s0100-879x2004000600001. Epub 2004 May 27. PMID 15264019
- [Background] Sperb F, Vairo F, Burin M, Mayer FQ, Matte U, Giugliani R. Genotypic and phenotypic characterization of Brazilian patients with GM1 gangliosidosis. Gene. 2013 Jan 1;512(1):113-6. doi: 10.1016/j.gene.2012.09.106. Epub 2012 Oct 6. PMID 23046582
- [Background] Caciotti A, Garman SC, Rivera-Colon Y, Procopio E, Catarzi S, Ferri L, Guido C, Martelli P, Parini R, Antuzzi D, Battini R, Sibilio M, Simonati A, Fontana E, Salviati A, Akinci G, Cereda C, Dionisi-Vici C, Deodato F, d'Amico A, d'Azzo A, Bertini E, Filocamo M, Scarpa M, di Rocco M, Tifft CJ, Ciani F, Gasperini S, Pasquini E, Guerrini R, Donati MA, Morrone A. GM1 gangliosidosis and Morquio B disease: an update on genetic alterations and clinical findings. Biochim Biophys Acta. 2011 Jul;1812(7):782-90. doi: 10.1016/j.bbadis.2011.03.018. Epub 2011 Apr 7. PMID 21497194
- [Background] Brunetti-Pierri N, Scaglia F. GM1 gangliosidosis: review of clinical, molecular, and therapeutic aspects. Mol Genet Metab. 2008 Aug;94(4):391-396. doi: 10.1016/j.ymgme.2008.04.012. Epub 2008 Jun 3. PMID 18524657
- [Background] Cachon-Gonzalez MB, Zaccariotto E, Cox TM. Genetics and Therapies for GM2 Gangliosidosis. Curr Gene Ther. 2018;18(2):68-89. doi: 10.2174/1566523218666180404162622. PMID 29618308
- [Derived] Ries M, Mendoza G, Arash-Kaps L, Amraoui Y, Quack F, Hardt B, Diederich S, Beck M, Mengel E. Quantitative longitudinal natural history of 8 gangliosidoses-conceptual framework and baseline data of the German 8-in-1 disease registry. A cross-sectional analysis. Genet Med. 2022 Dec;24(12):2434-2443. doi: 10.1016/j.gim.2022.09.001. Epub 2022 Oct 4. PMID 36194207